CLINICAL TRIAL: NCT06562153
Title: Tracking Brain Imaging Changes in Depression Over Clinical Accelerated Transcranial Magnetic Stimulation (TMS) Therapy at the Individual Level
Brief Title: fMRI Accelerated TMS Depression
Status: Recruiting | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Collaborators: Foundation for the Advancement of Clinical TMS (Unknown)
Responsible Party: Principal Investigator, Xiaolong Peng, Research Instructor, Medical University of South Carolina
Other Study IDs: Pro00138260
Record Dates: First submitted 2024-08-09; First posted 2024-08-20 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Depression
Keywords: Brain; Depression
MeSH Terms: conditions — Depression | interventions — Neuroimaging; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Volunteer Participants with Major Depressive Disorders (MDD): 20 patients with MDD receiving 5-day accelerated transcranial magnetic stimulation therapy (TMS) from the clinic will be recruited to participate in this observational neuroimaging study. Participants will undergo two fMRI scans at baseline and post-treatment.
  Interventions: Other: Neuroimaging with Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Other: Neuroimaging with Magnetic Resonance Imaging (MRI) — MRI will be used to observe brain states over time.

SUMMARY:
This study aims to investigate whether phenotypic-related brain states revealed by a novel INSCAPE ("Individualized Network-based Single-frame Coactivation Pattern Estimation") neuroimaging method in Major Depressive Disorder (MDD) patients can track brain recovery of MDD patients over an accelerated antidepressant transcranial magnetic stimulation (TMS) treatment.

DETAILED DESCRIPTION:
The aim of this study is to use magnetic resonance imaging (MRI) to capture images of participants' brains and apply an image processing method called INSCAPE to assess brain states. This study will recruit participants who are scheduled to receive accelerated Transcranial Magnetic Stimulation (TMS) therapy for Major Depressive Disorder (MDD). Participation in this study involves two visits, each including a 30-minute MRI scan. The interval between each visit is about one week. Depressed participants will also complete mood assessments at various intervals while they are receiving accelerated TMS for depression.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Have the capacity and ability to provide one's own consent in English and sign the informed consent document.
* DSM-IV diagnosis of MDD

Exclusion Criteria:

* Unable to speak English.
* Contraindicated for MRI.
* Any current or recent untreated medical, neurological, or psychiatric conditions
* Metal implant devices in the head, heart, or neck.
* History of brain surgery.
* History of cortisol medication use or electroconvulsive therapy.
* Comorbidity with other psychiatric/neurological illnesses or personality disorders
* History of myocardial infarction or arrhythmia, bradycardia.
* Personal history of head injury, concussion, or self-report of moderate to severe traumatic brain injury.
* Individuals suffering from frequent/severe headaches.
* Moderate to severe alcohol or substance use disorder.
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Volunteers with diagnosed MDD undergoing accelerated transcranial magnetic stimulation therapy (TMS).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2026-08-05 (Estimated); Study Completion 2026-08-05 (Estimated)

PRIMARY OUTCOMES:
Dynamic brain state change after 5-day transcranial magnetic stimulation (TMS) treatment compared to baseline | 5 days
  Two magnetic resonance imaging (MRI) scans will be collected at baseline and after the course of 5-day TMS treatment. A neuroimaging analysis method called "INSCAPE" will be used to get the dynamic brain state from the MRI data. The changes in brain states between baseline and after treatment MRI data will be calculated as the outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolong Peng, Principal Investigator — Medical University of South Carolina
Locations (1):
- 30 Bee Street, Charleston, South Carolina, United States